CLINICAL TRIAL: NCT00936702
Title: A Phase II Study of Carboplatin (CBDCA), Paclitaxel (TAXOL), and Everolimus (RAD001) in Previously Untreated Patients With Measurable Disease With Cancer of Unknown Primary (CUP)
Brief Title: Carboplatin, Paclitaxel, and Everolimus in Treating Patients With Previously Untreated Cancer of Unknown Primary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0871; NCI-2011-01926 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000643361 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma of Unknown Primary Origin
Keywords: Newly Diagnosed Carcinoma of Unknown Primary Origin; Squamous Cell Carcinoma of Unknown Primary Origin; Undifferentiated Carcinoma of Unknown Primary; newly diagnosed carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Carboplatin; Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carboplatin, paclitaxel, and everolimus) (Experimental): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Patients also receive everolimus PO QD on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: everolimus; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: everolimus — Given PO
Drug: paclitaxel — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well carboplatin given together with paclitaxel and everolimus works in treating patients with previously untreated cancer of unknown primary.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response rate in patients with previously untreated cancer of unknown primary treated with the combination of carboplatin, paclitaxel, and everolimus.

Secondary

* Assess time to progression, overall survival, duration of response, and time to treatment failure in patients treated with this regimen.
* Determine adverse events of this regimen in these patients.
* Perform descriptive correlative studies to determine response of specific tumor types, identified by the Origin-FFPE test, to this regimen.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Patients also receive oral everolimus once daily on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients' tumor tissue samples from the most recent biopsy are analyzed for correlative studies, including gene expression profiling by Origin-FFPE test.

After completion of study therapy, patients are followed up every 3 months until disease progression, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria

* Histological confirmation of metastatic adenocarcinoma, poorly differentiated non-small cell carcinoma, or poorly differentiated squamous carcinoma
* Adequate FFPE tissue or re-biopsy planned after registration but prior to treatment
* Measurable disease as defined; for patients having only lesions measuring at least 1 cm to =< 2 cm must use spiral computed tomography (CT) imaging for both pre- and post-treatment tumor assessments; disease that has received prior radiation (performed for palliative reasons) cannot be used for measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Hemoglobin (Hgb) >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet count >= 100,000/uL
* Total bilirubin =< upper limits of normal (ULN); if liver metastases are present, total bilirubin =< 2 x ULN
* Aspartate aminotransferase (AST) =< 2.5 x ULN; if liver metastases are present, AST =< 5 x ULN
* Creatinine =< 1.25 x ULN; if > 1.25 x ULN calculated creatinine clearance must be >= 60 ml/min
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willingness to return to NCCTG enrolling institution for follow-up
* Willingness to abstain from eating grapefruit or drinking grapefruit juice for the duration of the study

Exclusion Criteria

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception; note: adequate contraception must be used throughout the trial and for 8 weeks after the last dose of RAD001, by both sexes
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* History of any of the following:

  * Known to be human immunodeficiency virus (HIV) positive
  * Known prior/current history of hepatitis related to hepatitis B or hepatitis C
* Uncontrolled intercurrent illness including, but not limited to the following:

  * Ongoing or active infection (acute or chronic)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Severely impaired lung function
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN (note: optimal glycemic control should be achieved before starting trial therapy)
  * Liver disease such as cirrhosis or severe hepatic impairment
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 4 weeks prior to registration
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Untreated brain metastases; NOTE: patients with treated, stable brain metastases for at least 12 weeks prior to study entry are eligible for enrollment
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Active, bleeding diathesis
* Receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Currently on enzyme inducing anti-convulsants (EIACs) or other strong inducers or strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* Current use of warfarin (Coumadin); EXCEPTION: current use of low-molecular weight heparin is allowed
* Known to be HIV positive
* Inoculated with live attenuated vaccines =< 2 weeks prior to registration; note: close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus; examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* =< 4 weeks from major surgery; note: for this study, diagnostic laparoscopy (without other intervention) and/or biopsies (needle aspirate, core biopsy, open biopsy, etc.) are not considered major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, MD, Study Chair — Mayo Clinic
Locations (141):
- United States (141):
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Yoon HH, Foster NR, Meyers JP, Steen PD, Visscher DW, Pillai R, Prow DM, Reynolds CM, Marchello BT, Mowat RB, Mattar BI, Erlichman C, Goetz MP. Gene expression profiling identifies responsive patients with cancer of unknown primary treated with carboplatin, paclitaxel, and everolimus: NCCTG N0871 (alliance). Ann Oncol. 2016 Feb;27(2):339-44. doi: 10.1093/annonc/mdv543. Epub 2015 Nov 16. PMID 26578722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-six participants with centrally confirmed cancer of unknown primary site were enrolled between October 2009 and October 2012. The trial was closed before the target sample size of 50 was reached, because a sufficient number of confirmed responses had occurred to meet the primary endpoint.
Groups:
- Treatment (Carboplatin, Paclitaxel, and Everolimus): Patients receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Patients also receive everolimus PO QD on days 1, 8, and 15.
Period: Overall Study
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Started | 46
Completed | 0
Not Completed | 46
Not completed — Disease progression | 34
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 2
Not completed — Alternative Treatment | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 61 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 25
  1=Symptomatic and fully ambulatory | 15
  2=Symptomatic and ambulatory | 6
Histologic diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 36
  Poorly differentiated nonsmall-cell carcinoma | 5
  Poorly differentiated squamous carcinoma | 1
  Other | 4
Histologic grade [Count of Participants; unit: Participants]
  Well | 1
  Moderate | 8
  Poor | 28
  Undifferentiated, anaplastic | 8
  Not Available | 1
Predominant location of disease [Count of Participants; unit: Participants]
  Liver | 18
  Lung | 10
  Soft tissue | 9
  Bone | 3
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Tumor Responses
Description: Confirmed tumor response was defined to be either a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 4 weeks apart.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
Time Frame: First 6 Cycles of treatment (an average of 6 months)
Population: All participants except one who was deemed ineligible (treated prior to registration).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 45
percentage of participants | 36 [22 to 51]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from study enrollment to the time of death from any cause or last follow-up.
Time Frame: Time from registration to death or last follow-up (up to 3 years)
Population: All participants except one who was deemed ineligible (treated prior to registration).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 45
months | 10.1 [7.3 to 14.8]

3. Secondary Outcome: Progression-free Survival
Description: The progression-free survival (PFS) was defined as the time from date of registration to the documentation of disease progression or death as a result of any cause, whichever comes first.
Time Frame: Time from registration to the disease progression or death (up to 3 years)
Population: All participants except one who was deemed ineligible (treated prior to registration).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 45
months | 4.1 [2.8 to 5.7]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined for all evaluable participants who have achieved an objective response as the date at which the participant's objective status is first noted to be either CR or PR to the date progression is documented.
Time Frame: Up to 3 years
Population: All eligible participants who have achieved an objective response at which the participant's objective status is first noted to be either CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 16
months | 5.8 [2.5 to 6.8]

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined to be the time from the date of registration to the date at which the participant is removed from treatment due to progression, adverse events, or refusal.
Time Frame: Up to 3 years
Population: All participant who has been removed from treatment due to progression, adverse events, or refusal.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Number analyzed (Participants) | 40
months | 3.1 [1.6 to 4.2]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Treatment (Carboplatin, Paclitaxel, and Everolimus)
Serious Adverse Events (participants affected / at risk) | 21/46
Other Adverse Events (participants affected / at risk) | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carboplatin, Paclitaxel, and Everolimus) (N=46)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (8)
Cardiac disorder (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 15 (18)
Platelet count decreased (Investigations) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Carboplatin, Paclitaxel, and Everolimus) (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 44 (243)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Ascites (Gastrointestinal disorders) | 2 (6)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 21 (48)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 32 (93)
Vomiting (Gastrointestinal disorders) | 15 (25)
Edema limbs (General disorders) | 1 (3)
Fatigue (General disorders) | 20 (52)
Fever (General disorders) | 3 (4)
Pain (General disorders) | 2 (8)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 12 (15)
Bladder infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 4 (4)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 4 (10)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Forced expiratory volume decreased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 40 (205)
Lymphocyte count decreased (Investigations) | 3 (8)
Neutrophil count decreased (Investigations) | 38 (169)
Platelet count decreased (Investigations) | 31 (174)
Serum cholesterol increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 30 (93)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (10)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (5)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (46)
Seizure (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (73)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 17 (34)
Hypotension (Vascular disorders) | 1 (4)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less